CLINICAL TRIAL: NCT00927394
Title: An 8 Week Randomized, Double-Blind, Parallel Group, Multi-Center, Active Controlled Study to Evaluate the Antihypertensive Efficacy and Safety of Aliskiren Administered in Combination With Valsartan Versus Valsartan Alone in Patients With Stage 2 Systolic Hypertension and Type 2 Diabetes Mellitus
Brief Title: Aliskiren and Valsartan vs Valsartan Alone in Patients With Stage II Systolic Hypertension and Type II Diabetes Mellitus
Acronym: ViVID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPV100AUS02
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Hypertension
Keywords: Hypertension, Type II Diabetes, Aliskiren, Valsartan,; Systolic blood pressure, Diastolic blood pressure,; Stage II, Combination
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — aliskiren; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Combination Therapy: Aliskiren + Valsartan (Experimental): To adequately blind the study, patients were required to take a total of 4 tablets/capsules a day (2 tablets and 2 capsules of study drug per day)for 8 weeks. 1 tablet of Aliskiren 150 mg + 1 tablet of placebo Aliskiren 150 mg + 1 capsule of Valsartan 160 mg + 1 capsule of placebo Valsartan 160 mg daily for 2 weeks. Forced titrated to: 2 tablets of Aliskiren 150 mg + 2 capsules of Valsartan 160 mg daily for 6 weeks
  Interventions: Drug: Aliskiren; Drug: Valsartan; Drug: Placebo for Aliskiren; Drug: Placebo for Valsartan
- Monotherapy: Valsartan (Active Comparator): To adequately blind the study, patients were required to take a total of 4 tablets/capsules a day (2 tablets and 2 capsules of study drug per day) for 8 weeks. 1 capsule of Valsartan 160 mg + 1 capsule of placebo Valsartan 160 mg + 2 tablets of placebo Aliskiren 150 mg daily for 2 weeks. Forced titrated to: 2 capsules of Valsartan 160 mg + 2 tablets of placebo Aliskiren 150 mg daily for 6 weeks.
  Interventions: Drug: Valsartan; Drug: Placebo for Aliskiren; Drug: Placebo for Valsartan

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150 mg tablet
  Arms: Combination Therapy: Aliskiren + Valsartan
Drug: Valsartan — Valsartan 160 mg capsules
Drug: Placebo for Aliskiren — Placebo for Aliskiren 150 mg tablets
Drug: Placebo for Valsartan — Placebo for Valsartan 160 mg capsules

SUMMARY:
The purpose of the study was to evaluate the blood pressure (BP)-lowering efficacy of the combination of aliskiren and valsartan, as initial therapy, compared to valsartan monotherapy in Type II Diabetic patients with Stage II hypertension.

DETAILED DESCRIPTION:
When protocol Amendment 2 was released, there were patients who had already been randomized into the study. These patients were included in the trial prior to making changes to the eligibility criteria. Thus, the study contains 2 distinct cohorts. Cohort 1 contains those patients who had already been randomized, and had been deemed eligible based on the original inclusion/exclusion criteria, prior to Amendment 2. No new patients were randomized to Cohort 1. Cohort 2 contains patients who were randomized, having been found eligible based on the revised inclusion/exclusion criteria, after Amendment 2. Differences in the inclusion and exclusion criteria are indicated below.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible and able to participate in the study, and who give written informed consent before any assessment is performed.
* Men or women 18 years and older.
* Patients with Type 2 diabetes mellitus with an HbA1c ≤ 9 % at visit 1 and on a stable anti-diabetic regimen not including insulin or stable diet and exercise for at least 4 weeks prior to visit 1.

Cohort 1:

* Patients with Stage 2 systolic hypertension, defined as having a MSSBP ≥160 mmHg and <200 mmHg at Visit 5 (randomization).
* Patients who have been newly diagnosed with hypertension or who have not received antihypertensive medication for at least 4 weeks (28 days) prior to Visit 1 must have MSSBP ≥ 160 mmHg and < 200 mmHg at Visit 1, otherwise, they will be considered screen failures.
* Patients receiving antihypertensive medication must have a MSSBP of ≥150 mmHg and <200 mmHg at Study Visit 1, otherwise they will be considered screen failures.

Cohort 2:

* Patients must also have had a mean 8-hour daytime ambulatory systolic blood pressure (ASBP) ≥140 mmHg AND mean 8-hour daytime ambulatory diastolic blood pressure (ADBP) ≥90 mmHg at Visit 5 (randomization).
* Hypertensive patients with MSSBP ≥150 mmHg and but <200 mmHg AND MSDBP ≥95 but <120 mmHg at Visit 5 (randomization).
* Patients who had been newly diagnosed with hypertension or who had not received antihypertensive medication for at least 4 weeks (28 days) prior to Visit 1 must have had MSSBP ≥150 mmHg but <200 mmHg and MSDBP ≥95 but <120 mmHg at Visit 1, otherwise, they were considered screen failures.

Exclusion Criteria:

* Office blood pressure measured by cuff (MSSBP ≥200 mmHg or MSDBP ≥120 mmHg).
* History or evidence of secondary hypertension of any etiology.
* Refractory hypertension, defined as having uncontrolled BP (≥140/90 mmHg) while receiving 3 antihypertensive medications at the maximum approved dose of each drug, one of which must be a diuretic.
* Patients treated with more than 3 antihypertensive medications (each component of a combination drug counts individually).
* Type 2 diabetes mellitus currently requiring insulin treatment.
* modification of diet in renal disease (MDRD) estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2
* Serum sodium less than lower limit of normal, serum potassium < 3.5 mEq/L or ≥ 5.3 mEq/L at Visit 1.
* Known Keith-Wagener grade III or IV hypertensive retinopathy.

Cohort 1:

- Patients with known diabetic retinopathy (eg, having a history of laser therapy for diabetic retinopathy) or diabetic neuropathy (eg, receiving medication for diabetic neuropathy).

Cohort 2:

- Patients with known diabetic retinopathy or diabetic neuropathy and/or having a history of treatment for either.

Other protocol-defined inclusion/exclusion criteria applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1143 (Actual)
Dates: Start 2009-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (4):
- United States (4):
  - Investigative Site, Newark, Delaware
  - Investigative Site, Kansas City, Missouri
  - Investigative Site, Camden, New Jersey
  - Investigative Site, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Bakris GL, Oparil S, Purkayastha D, Yadao AM, Alessi T, Sowers JR. Randomized study of antihypertensive efficacy and safety of combination aliskiren/valsartan vs valsartan monotherapy in hypertensive participants with type 2 diabetes mellitus. J Clin Hypertens (Greenwich). 2013 Feb;15(2):92-100. doi: 10.1111/jch.12032. Epub 2012 Oct 26. PMID 23339726

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Started | 575 | 568 (One patient was randomized in error and was discontinued by site.)
Cohort 1 (Randomized) | 157 (Cohort 1 includes patients with specific eligibility criteria mentioned in protocol section) | 165
Cohort 2 (Randomized) | 418 (Cohort 2 includes patients with specific eligibility criteria mentioned in protocol section) | 403
Combined Safety Set (Cohort 1 and 2) | 574 | 565
Cohort 1: Full Analysis Set 1 (FAS 1) | 157 (FAS 1 includes all patients in Cohort 1 to whom study treatments were given through randomization.) | 164
Cohort 2: Full Analysis Set 2 (FAS 2) | 417 (FAS 2= all patients randomized to Cohort 2 and who had a valid baseline assessment of 24 hours ABPM.) | 398
FAS 2 :Ambulatory Blood Pressure Monitor | 342 (consists of all patients in FAS 2 who had both valid baseline and post-baseline ABPM assessments.) | 323
Combined Full Analysis Set (FAS 1+FAS 2) | 574 | 562
Completed | 498 | 483
Not Completed | 77 | 85
Not completed — Adverse Event | 14 | 9
Not completed — Unsatisfactory therapeutic effect | 17 | 23
Not completed — Withdrawal by Subject | 20 | 24
Not completed — Lost to Follow-up | 8 | 14
Not completed — Administrative Problem | 1 | 0
Not completed — Death | 1 | 1
Not completed — Protocol deviation | 16 | 13
Not completed — Randomized in error | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan | Total
Number analyzed (Participants) | 574 | 565 | 1139
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic measures were based on Safety set.
  years | 55.0 (9.30) | 55.2 (9.60) | 55.1 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 244 | 477
  Male | 341 | 321 | 662

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean 24-hour Ambulatory Systolic Blood Pressure (MASBP) at Week 8
Description: The 24-hour ambulatory systolic blood pressure was evaluated at baseline (Week 0) and post-baseline visits. The mean hourly systolic blood pressure was calculated at post-dosing hours 1-24 for each patient. The MASBP for each patient was calculated by averaging the patient's available hourly means for post-dosing hours 1-24.
Time Frame: baseline, week 8
Population: Full Analysis Set 2 (FAS 2) with ambulatory blood pressure monitoring (ABPM)- Consists of all patients in Cohort 2 to whom study treatments were assigned through randomization and who had both valid baseline and post-baseline ambulatory blood pressure monitoring (ABPM)assessments.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Number analyzed (Participants) | 342 | 323
mmHg | -15.3 (14.62) | -11.5 (14.75)

2. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (MSSBP)
Description: Sitting blood pressure was measured at trough (24 hours ± 3 hours post dose) and recorded at all study visits. At the first study visit, the arm in which the highest sitting diastolic blood pressure was found was the arm used for all subsequent readings throughout the study. At each study visit, after the patient had been sitting for five minutes, systolic and diastolic blood pressures were measured 3 times using the standard mercury sphygmomanometer. The repeat sitting measurements were made at 1-2 minute intervals and the mean of these 3 sitting blood pressure measurements was used as the average sitting office blood pressure for that visit.
Time Frame: Baseline, week 8
Population: Combined FAS included all randomized patients in Cohort 1 (FAS 1) and all randomized patients in Cohort 2 who had a valid baseline assessment of 24-hour ambulatory systolic blood pressure measurement (FAS 2). Patients with baseline and week 8 data were included in this analysis. Last-observation-carried-forward (LOCF) approach was used.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Combination Therapy: Aliskiren + Valsartan: To adequately blind the study, patients were required to take a total of 4 tablets/capsules a day (2 tablets and 2 capsules of study drug per day) for 8 weeks. 1 tablet of Aliskiren 150 mg + 1 tablet of placebo Aliskiren 150 mg + 1 capsule of Valsartan 160 mg + 1 capsule of placebo Valsartan 160 mg daily for 2 weeks. Forced titrated to: 2 tablets of Aliskiren 150 mg + 2 capsules of Valsartan 160 mg daily for 6 weeks
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Number analyzed (Participants) | 562 | 553
mmHg | -21.7 (18.70) | -18.2 (18.06)

3. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory Diastolic Blood Pressure (MADBP) at Week 8
Description: The 24-hour ambulatory diastolic blood pressure was evaluated at baseline (Week 0) and post-baseline visits. The mean hourly diastolic blood pressure was calculated at post-dosing hours 1-24 for each patient. The MADBP for each patient was calculated by averaging the patient's available hourly means for post-dosing hours 1-24.
Time Frame: baseline, week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Number analyzed (Participants) | 342 | 323
mmHg | -9.2 (8.80) | -6.7 (8.82)

4. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory Pulse Pressure (MAPP) at Week 8
Description: The 24-hour ambulatory pulse pressure was evaluated at baseline (Week 0) and post-baseline visits.
Time Frame: baseline, week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Number analyzed (Participants) | 342 | 323
mmHg | -6.1 (8.58) | -4.7 (8.26)

5. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (MSDBP)
Description: as for outcome 2
Time Frame: Baseline, week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Number analyzed (Participants) | 562 | 553
mmHg | -11.0 (10.58) | -8.3 (10.60)

6. Secondary Outcome: Change From Baseline in Mean Sitting Pulse Pressure (MSPP) at Week 8
Description: At each visit, the pulse rate was measured for 30 seconds just prior to the first sitting blood pressure measurement.
Time Frame: baseline, week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Number analyzed (Participants) | 562 | 553
mmHg | -10.8 (13.46) | -9.9 (13.83)

7. Secondary Outcome: Percentage of Patients Achieving Blood Pressure Control
Description: Blood pressure control was defined as MSSBP/MSDBP <140/90 mmHg. Percentage of patients achieving of blood pressure control at the corresponding visit was reported
Time Frame: 8 weeks
Population: Combined FAS included all randomized patients in Cohort 1 (FAS 1) and all randomized patients in Cohort 2 who had a valid baseline assessment of 24-hour ambulatory systolic blood pressure measurement (FAS 2). Number of patients with data at each visit were analyzed.
Measure: Number; unit: Percentage of patients
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Number analyzed (Participants) | 514 | 498
Percentage of patients | 39.9 | 32.7

8. Secondary Outcome: Percentage of Responders
Description: Responders were defined as patients with MSSBP <130 mmHg or a reduction from baseline in MSSBP of >20 mmHg.Percentage of responders achieving a response at the corresponding visit was reported.
Time Frame: Baseline, Week 8
Population: Combined FAS included all randomized patients in Cohort 1 (FAS 1) and all randomized patients in Cohort 2 who had a valid baseline assessment of 24-hour ambulatory systolic blood pressure measurement (FAS 2). Patients with baseline and week 8 assessments were included in this analysis.
Measure: Number; unit: Percentage of patients
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Number analyzed (Participants) | 514 | 498
Percentage of patients | 61.9 | 53.8

9. Secondary Outcome: Change From Baseline in Plasma Renin Activity (PRA) at Week 8
Time Frame: Baseline, week 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL/hr
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Number analyzed (Participants) | 429 | 409
ng/mL/hr | 1.056 (4.966) | 0.879 (4.646)

10. Secondary Outcome: Change From Baseline in Plasma Renin Concentration (PRC) at Week 8
Time Frame: Baseline, week 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Number analyzed (Participants) | 428 | 404
ng/L | 68.592 (209.544) | 124.721 (489.719)

11. Secondary Outcome: Change From Baseline in Plasma Aldosterone at Week 8
Time Frame: Baseline, week 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Number analyzed (Participants) | 431 | 411
pmol/L | -21.957 (115.251) | -22.562 (123.343)

12. Secondary Outcome: Number of Patients With Adverse Events, Serious Adverse Events and Death
Description: Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen.
  Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: 8 weeks
Population: Safety Set - Consisted of all patients who received at least one dose of double-blind trial medication. Patients were analyzed according to the treatment that they received.
Measure: Number; unit: Patients
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Number analyzed (Participants) | 574 | 565
Patients
  Adverse Events | 202 | 182
  Serious Adverse events | 9 | 9
  Death | 1 | 1

ADVERSE EVENTS:
Description: Safety Set - Consists of all patients who received at least one dose of double-blind trial medication. Patients were analyzed according to the treatment that they received.
Arm/Group | Combination Therapy: Aliskiren + Valsartan | Monotherapy: Valsartan
Serious Adverse Events (participants affected / at risk) | 9/574 | 9/565
Other Adverse Events (participants affected / at risk) | 34/574 | 36/565
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy: Aliskiren + Valsartan (N=574) | Monotherapy: Valsartan (N=565)
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Sweat gland infection (Infections and infestations) | 0 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy: Aliskiren + Valsartan (N=574) | Monotherapy: Valsartan (N=565)
Headache (Nervous system disorders) | 34 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.